CLINICAL TRIAL: NCT00297206
Title: An Open-label, Single-dose, Multicenter, Pharmacokinetic, Safety and Tolerability Study of Valaciclovir Oral Suspension in Infants and Children.
Brief Title: A Safety And Tolerability Study Of Valaciclovir Oral Suspension In Infants And Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS210914
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Herpes Simplex
Keywords: pharmacokinetics herpes varicella herpes labialis Epstein-Barr virus
MeSH Terms: conditions — Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Subjects in the age group of 2 to less than 6 years will be included
  Interventions: Drug: Valaciclovir
- Cohort 2 (Experimental): Subjects in the age group of 1 to less than 2 years will be included
  Interventions: Drug: Valaciclovir
- Cohort 3 (Experimental): Subjects in the age group of 6 months to less than 1 year will be included
  Interventions: Drug: Valaciclovir
- Cohort 4 (Experimental): Subjects in the age group of 3 months to less than 6 months will be included
  Interventions: Drug: Valaciclovir
- Cohort 5 (Experimental): Subjects in the age group of 1 month to less than 3 months will be included
  Interventions: Drug: Valaciclovir

INTERVENTIONS:
Drug: Valaciclovir — Valaciclovir will be administered as an extemporaneously prepared suspension formulation. Valaciclovir oral suspension will be prepared by crushing marketed Valtrex Caplets 500 milligram (mg) and suspending the resultant powder in Suspension Structured Vehicle USNF with dose strength of 25 milligram per milliliter (mg/mL) or 50 mg/mL.

SUMMARY:
Limited data are available on valaciclovir use in children and valaciclovir is not currently approved for use in pediatrics. The marketed formulation of valaciclovir is not ideal for use in pre-adolescent patients who may have trouble swallowing solid oral dosage forms. An extemporaneous suspension formulation of valaciclovir has been developed to expedite the provision of benefits to children similar to those from administration of valaciclovir solid formulations in adults.

ELIGIBILITY:
Inclusion criteria:

* Subjects who have a current herpes virus infection.
* Have neonatally acquired herpes at risk of potential recurrence.
* Immunocompromised or cancer patients at risk for development of a herpes virus infection.

Exclusion criteria:

* Hypersensitivity to antiherpetic medications.
* Impaired hepatic or renal function.
* Show presence of other serious or unstable underlying disease.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2003-01-25 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2007-02-28 (Actual)

PRIMARY OUTCOMES:
Plasma acyclovir and valaciclovir concentrations pre-dose (within 15 minutes of dose administration) and at 0.5, 1, 2, 4 and 6 hours following administration of the valaciclovir oral suspension dose. | 0.5, 1, 2, 4 and 6 hours

SECONDARY OUTCOMES:
Safety monitoring throughout the study and at the follow up evaluation 2-4 days after the single dose of study medication. | Up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (10):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Galveston, Texas
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- South Africa (2):
  - GSK Investigational Site, Brits
  - GSK Investigational Site, George

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bradley J, Scholtz F, Brennan C, Zhao H, Weller S. Pharmacokinetics and safety of single-dose valacyclovir oral suspension in infants and children with current or potential herpesvirus infection. Poster presentation, 45th Annual Meeting Infectious Disease
- [Background] Kimberlin DW, Jacobs RF, Weller S, van der Walt JS, Heitman CK, Man CY, Bradley JS. Pharmacokinetics and safety of extemporaneously compounded valacyclovir oral suspension in pediatric patients from 1 month through 11 years of age. Clin Infect Dis. 2010 Jan 15;50(2):221-8. doi: 10.1086/649212. PMID 20014952
- See also: Results for study HS210914 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/HS210914?search=study&search_terms=HS210914#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HS210914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register